CLINICAL TRIAL: NCT00580996
Title: Water and the Gastropressor Response - Tachyphylaxis (Specific Aim 1.2)
Brief Title: Water and the Gastropressor Response - Tachyphylaxis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Satish R. Raj (Other)
Responsible Party: Sponsor-Investigator, Satish R. Raj, Assistant Professor of Medicine & Pharmacology, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 060547; Vanderbilt Discovery (Other: Vanderbilt Univeristy)
Record Dates: First submitted 2007-12-22; First posted 2007-12-27 (Estimated); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Orthostatic Hypotension
Keywords: water; orthostatic hypotension; blood pressure
MeSH Terms: conditions — Hypotension, Orthostatic | interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 16 oz water in AM
  Interventions: Other: water high dose
- 2 (Active Comparator): water 1 oz in AM
  Interventions: Other: water tiny dose

INTERVENTIONS:
Other: water high dose — water 16 oz PO x 1
  Arms: 1
Other: water tiny dose — water 1 oz PO x 1
  Arms: 2

SUMMARY:
We are studying the effects of oral water ingestion in patients with orthostatic hypotension. In this study, we are testing the null hypothesis that the blood pressure increase with oral water ingestion will not be diminished if a full prior water dose is given a few hours earlier.

DETAILED DESCRIPTION:
We are studying the effects of oral water ingestion in patients with orthostatic hypotension. This has been termed the Gastropressor Response. In this study, we are testing the null hypothesis that the blood pressure increase with oral water ingestion will not be diminished if a full prior water dose is given a few hours earlier. In this 2 day study, subjects will be asked to drink with 1 oz or 16 oz of water in the morning followed a few hours later by 16 oz water while the blood pressure is monitored. On the 2nd day, the other dose of water will be given to start, with 16 oz again as the second dose.

ELIGIBILITY:
Inclusion Criteria:

* orthostatic hypotension (fall in BP>20/10 mmHg)
* pressor response to water in other studies
* Age 18-80 years

Exclusion Criteria:

* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-07; Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
blood pressure | 2nd water intervention

SECONDARY OUTCOMES:
heart rate | 2nd intervention

CONTACTS AND LOCATIONS:
Overall Officials: Satish R Raj, MD MSCI, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt Autonomic Dysfunction Center website — https://www.vumc.org/autonomic-dysfunction-center/vanderbilt-autonomic-dysfunction